CLINICAL TRIAL: NCT04628117
Title: Assess Effect of Oral Nutritional Supplementation on Oxidative Stress Levels in Protein-energy Wasting Patients With Continuous Ambulatory Peritoneal Dialysis
Brief Title: Effect of Oral Nutritional Supplementation on Oxidative Stress in Protein-energy Wasting Patients With Peritoneal Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Civil Juan I. Menchaca (Other)
Responsible Party: Principal Investigator, Francisco Gerardo Yanowsky Escatell, Principal Investigator, Hospital Civil Juan I. Menchaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HospitalCJIM
Record Dates: First submitted 2020-10-28; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Oxidative Stress; Protein-Energy Wasting; Malnutrition; Protein-Energy Malnutrition; Oral Nutritional Supplements; Peritoneal Dialysis
MeSH Terms: conditions — Malnutrition; Protein-Energy Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with two-parallel-group in stable continuous ambulatory peritoneal dialysis patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Nutritional counselling by individualized nutritional plan for 8 weeks.
- Oral nutritional supplementation (Experimental): Nutritional counselling by individualized nutritional plan plus oral nutritional supplementation for renal disease (237 mls per day) for 8 weeks.
  Interventions: Dietary Supplement: Oral nutritional supplementation for kidney disease

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplementation for kidney disease — 237 mls per day for 8 weeks.
  Arms: Oral nutritional supplementation

SUMMARY:
End-stage kidney disease (ESKD) represents a serious public health problem in Mexico. Data from the United States Renal Data System (USRDS) have reported that the region of Jalisco (Mexico) is one of the places with the highest incidence rate of treated ESKD and use of peritoneal dialysis (PD). In patients with ESKD, oxidative stress (OS) has been recognized as a potential source of morbidity and mortality, since it is involved in the pathogenesis of atherosclerosis and other complications of ESRD. This can induce damage to DNA (nucleic acid), proteins, carbohydrates, and lipids.

Another common complication in ESKD patients receiving PD is protein-energy wasting (PEW), which is characterized by the decline in the body stores of protein and energy fuels (that is, body protein and fat masses) due to the multiple nutritional and catabolic alterations that occur in this condition. Diverse factors can affect the nutritional and metabolic status of patients with PD, for which they require interventions to reverse protein and energy depletion. Nutritional counseling can be a useful tool in PD patients in order to improve compliance with nutritional recommendations. The strategies more used for PEW include oral nutritional supplementation. Therefore, the purpose of this study is assess the effect of oral nutritional supplementation on OS in PEW patients with PD.

DETAILED DESCRIPTION:
The detection of patients is carried out in the Nephrology Service of the Hospital Civil de Guadalajara Dr. Juan I. Menchaca where the selection and exclusion criteria are evaluated.

The probabilistic group assignment is carried out using a sealed and opaque envelope.

Control group: only nutritional counselling for 8 weeks. Intervention group: nutritional counselling plus 237 mls per day of oral nutritional supplement for kidney disease.

Initial evaluation includes, anthropometric parameters and dietary intake. Demographic characteristics and OS levels, such as oxidants, antioxidants and oxidative DNA damage.

All nutritional counselling, dietary intake, medical nutrition theraphy (oral nutritional supplementation), assessment of OS levels, and anthropometric parameters will perform at 0, 4 and 8 weeks of follow up. Protein-energy wasting assessment only in the 0 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of protein-energy wasting evaluated by 7-point Subjective Global Assessment (moderate/severe), and Malnutrition-inflammation Score (a score ≥ 6).
* Male and female patients
* Age ≥ 18 and <60 years
* Receive continuous ambulatory peritoneal dialysis with at least 3 months of initiation of renal replacement therapy
* Patients without clinical or biochemical evidence of any infectious process (peritonitis, urosepsis, endocarditis, soft tissue infection, pneumonia, etc) or inflammatory systemic disease (systemic lupus erythematosus, vasculitis, connective tissue disease)
* Written informed consent

Exclusion Criteria:

* Supplementation with exogenous antioxidants 2 months prior
* Smoking less than 1 year
* Intermittent peritoneal dialysis or automated peritoneal dialysis
* PD catheter dysfunction
* Known allergy or intolerance to oral nutritional supplement for renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-10-04 (Estimated); Primary Completion 2022-05-28 (Estimated); Study Completion 2023-03-11 (Estimated)

PRIMARY OUTCOMES:
Change in oxidative stress levels, oxidants (products of Lipoperoxidation, 8-IP, NO), antioxidants (SOD, catalase, GPx, TAC), and oxidative DNA damage (8-OHdG, hOGG1). | 8 weeks
  As measured by the of OS markers, 10 mL of blood samples will be taken prior to nutritional evaluation, 5 mL with 0.1% of ethylenediaminetetraacetic (EDTA) tube and other 5 mL in dry tube. The blood will be centrifuged at 10,000 rpm for 10 min at room temperature; supernatants were stored in aliquots at -80°C until its final processing.

SECONDARY OUTCOMES:
Change protein-energy wasting and dietary intake | 8 weeks
  Description: As measured by 7-point Subjective Global Assesment (SGA), SGA of 1-2 for severe PEW, 3-5 for mild-moderate protein energy wasting will be considered as presence of protein-energy wasting and malnutrition inflammation score (MIS) a score ≥ 6 will be considered as the presence of protein-energy wasting.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sung CC, Hsu YC, Chen CC, Lin YF, Wu CC. Oxidative stress and nucleic acid oxidation in patients with chronic kidney disease. Oxid Med Cell Longev. 2013;2013:301982. doi: 10.1155/2013/301982. Epub 2013 Aug 24. PMID 24058721
- [Background] Liakopoulos V, Roumeliotis S, Gorny X, Eleftheriadis T, Mertens PR. Oxidative Stress in Patients Undergoing Peritoneal Dialysis: A Current Review of the Literature. Oxid Med Cell Longev. 2017 Dec 27;2017:3494867. doi: 10.1155/2017/3494867. eCollection 2017. PMID 29750088
- [Background] Roumeliotis S, Eleftheriadis T, Liakopoulos V. Is oxidative stress an issue in peritoneal dialysis? Semin Dial. 2019 Sep;32(5):463-466. doi: 10.1111/sdi.12818. Epub 2019 May 1. PMID 31044475
- [Background] Kochlik B, Grune T, Weber D. New findings of oxidative stress biomarkers in nutritional research. Curr Opin Clin Nutr Metab Care. 2017 Sep;20(5):349-359. doi: 10.1097/MCO.0000000000000388. PMID 28562491
- [Background] Domenici FA, Vannucchi MT, Jordao AA Jr, Meirelles MS, Vannucchi H. DNA oxidative damage in patients with dialysis treatment. Ren Fail. 2005;27(6):689-94. doi: 10.1080/08860220500242678. PMID 16350819
- [Background] Fouque D, Kalantar-Zadeh K, Kopple J, Cano N, Chauveau P, Cuppari L, Franch H, Guarnieri G, Ikizler TA, Kaysen G, Lindholm B, Massy Z, Mitch W, Pineda E, Stenvinkel P, Trevino-Becerra A, Wanner C. A proposed nomenclature and diagnostic criteria for protein-energy wasting in acute and chronic kidney disease. Kidney Int. 2008 Feb;73(4):391-8. doi: 10.1038/sj.ki.5002585. Epub 2007 Dec 19. PMID 18094682
- [Background] Carrero JJ, Stenvinkel P, Cuppari L, Ikizler TA, Kalantar-Zadeh K, Kaysen G, Mitch WE, Price SR, Wanner C, Wang AY, ter Wee P, Franch HA. Etiology of the protein-energy wasting syndrome in chronic kidney disease: a consensus statement from the International Society of Renal Nutrition and Metabolism (ISRNM). J Ren Nutr. 2013 Mar;23(2):77-90. doi: 10.1053/j.jrn.2013.01.001. PMID 23428357
- [Background] Ikizler TA, Cano NJ, Franch H, Fouque D, Himmelfarb J, Kalantar-Zadeh K, Kuhlmann MK, Stenvinkel P, TerWee P, Teta D, Wang AY, Wanner C; International Society of Renal Nutrition and Metabolism. Prevention and treatment of protein energy wasting in chronic kidney disease patients: a consensus statement by the International Society of Renal Nutrition and Metabolism. Kidney Int. 2013 Dec;84(6):1096-107. doi: 10.1038/ki.2013.147. Epub 2013 May 22. PMID 23698226
- [Background] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133
- [Background] Prasad N, Gupta A, Sinha A, Sharma RK, Kumar A, Kumar R. Changes in nutritional status on follow-up of an incident cohort of continuous ambulatory peritoneal dialysis patients. J Ren Nutr. 2008 Mar;18(2):195-201. doi: 10.1053/j.jrn.2007.08.002. PMID 18267212
- [Background] Martin-Del-Campo F, Gonzalez-Espinoza L, Rojas-Campos E, Ruiz N, Gonzalez J, Pazarin L, Cueto-Manzano AM. Conventional nutritional counselling maintains nutritional status of patients on continuous ambulatory peritoneal dialysis in spite of systemic inflammation and decrease of residual renal function. Nephrology (Carlton). 2009 Aug;14(5):493-8. doi: 10.1111/j.1440-1797.2008.01081.x. PMID 19674317
- [Background] Ikizler TA, Burrowes JD, Byham-Gray LD, Campbell KL, Carrero JJ, Chan W, Fouque D, Friedman AN, Ghaddar S, Goldstein-Fuchs DJ, Kaysen GA, Kopple JD, Teta D, Yee-Moon Wang A, Cuppari L. KDOQI Clinical Practice Guideline for Nutrition in CKD: 2020 Update. Am J Kidney Dis. 2020 Sep;76(3 Suppl 1):S1-S107. doi: 10.1053/j.ajkd.2020.05.006. PMID 32829751